CLINICAL TRIAL: NCT06728878
Title: Lymph Node Metastasis and Tumor Deposit in the Short Gastric Mesentery Following Total Gastrectomy With D2 Lymphadenectomy Plus Complete Mesogastric Excision for Gastric Cancer: A Prospective Observational Study
Brief Title: Analysis of Lymph Node Metastasis and Tumor Deposit in the Short Gastric Mesentery Following Total Gastrectomy for Gastric Cancer
Acronym: zytg001
Status: Recruiting | Type: Observational
Sponsor: Jichao Qin (Other)
Responsible Party: Sponsor-Investigator, Jichao Qin, Professor, First Affiliated Hospital of Zhejiang University
Organization: First Affiliated Hospital of Zhejiang University (Other)
Other Study IDs: 2024-0899-1
Record Dates: First submitted 2024-09-01; First posted 2024-12-11 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Gastric Cancers
Keywords: Gastric cancer; Lymph node dissection; Short gastric mesentery; Lymph node metastasis; Tumor location
MeSH Terms: conditions — Stomach Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients who received total gastrectomy with D2 lymphadenectomy plus complete mesogastric excision: No additional intervention is imposed on patients except normal clinical diagnosis and treatment.

SUMMARY:
This study aims to explore lymph node metastasis in the short gastric mesentery following total gastrectomy with D2 lymphadenectomy plus complete mesogastric excision, providing evidence-based medicine for standardizing lymph node dissection in gastric cancer.

DETAILED DESCRIPTION:
According to the 6th edition of the Japanese Gastric Cancer Treatment Guidelines; total gastrectomy with D2 lymphadenectomy includes groups No.1 to No.7, No.8a, No.9, No.11p, No.11d, and No.12a. The No.4sa group lymph nodes are defined as the lymph nodes along the short gastric vessel, No.10 group lymph nodes are defined as the lymph nodes at the splenic hilum including the lymph nodes at the roots of the short gastric arteries. In routine total gastrectomy with D2 combined with CME surgery, the standard practice involves resection of the short gastric mesentery (No.4sa group and No. 10 group). There are typically 3-4 short gastric arteries in the human body, further investigation is required to determine the lymph node metastasis rates in each short gastric mesentery. Patients undergoing total gastrectomy with D2 combined with CME will have their short gastric mesenteries anatomically separated for examination, and this aims to analyze the positive rate of lymph nodes in the short gastric mesentery and investigate the correlation between tumor location, staging, and lymph node metastasis in the short gastric mesentery.

ELIGIBILITY:
Inclusion Criteria:

1. Aged older than 18 years and younger than 85 years
2. Primary gastric adenocarcinoma confirmed by preoperative pathology result
3. cT2-4aN0-3M0 at preoperative evaluation according to the American Joint 8 Committee on Cancer (AJCC) Cancer Staging Manual 8th Edition
4. Patients who received total gastrectomy with D2 lymphadenectomy plus complete mesogastric excision
5. American Society of Anesthesiologists (ASA) class I, II, or III
6. Written informed consent

Exclusion Criteria:

1. Negative preoperative biopsy
2. Too late tumour stage or metastasis (cT4b/M1)
3. BMI>30 kg/m2
4. previous neoadjuvant chemotherapy or radiotherapy
5. Previous upper abdominal surgery
6. Combined with other malignant diseases
7. Reject operation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received total gastrectomy with D2 lymphadenectomy plus complete mesogastric excision. At the same time, the patients met the above inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of lymph node metastasis and tumor deposit in the short gastric mesentery | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastrointestinal Surgery, The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided